CLINICAL TRIAL: NCT04154475
Title: Dairy Intervention in People With Obesity
Acronym: DIPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIPO 1.0
Record Dates: First submitted 2019-10-16; First posted 2019-11-06 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Obesity
Keywords: yogurt; dairy; calcium; weight reduction; obesity; randomized controlled trial; body composition; microbiome
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- yogurt diet (Experimental): yogurt-diet (-500 kcal/day, 500 g yogurt, high calcium)
  Interventions: Dietary Supplement: yogurt diet
- dairy diet (Active Comparator): dairy diet: -500 kcal/day, high calcium, 500 g non-yogurt dairy products
  Interventions: Dietary Supplement: dairy diet
- standard diet (Active Comparator): standard diet: -500 kcal/day, low calcium, 500 g soya-yogurt
  Interventions: Dietary Supplement: standard diet

INTERVENTIONS:
Dietary Supplement: yogurt diet — 500 g yogurt/day
  Arms: yogurt diet
Dietary Supplement: dairy diet — 500 g non-yogurt dairy products
  Arms: dairy diet
Dietary Supplement: standard diet — 500 g soya-yogurt
  Arms: standard diet

SUMMARY:
Obesity is associated with increased morbidity and mortality, but weight reduction is difficult to achieve. In this randomized controlled trial we will include 120 obese subjects. Subjects will be allocated to one of the 3 diet types (minus 500 kcal / d):

* Yoghurt diet: 500 g low-fat yogurt / d, about 1000-1100 mg calcium / d,
* Milk product diet: 500 g of low-fat milk or buttermilk / d, about 1000-1100 mg calcium / d
* Standard diet: 500 g soy yogurt / d, about 500 mg calcium / d Primary endpoint is the change in fat mass (baseline vs. 12 weeks), secondary endpoints are metabolic and endocrine parameters, gut microbiome, quality of life, hunger and satiety.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30 kg/m²
* Age of ≥18 and <60 years
* Written informed consent before study entry
* Willingness to introduce a dietary change to lose weight

Exclusion Criteria:

* Serum calcium ≥2.7 mmol/l
* Dislike or intolerance of dairy products, reporting adverse responses or allergy to dairy products
* Pregnancy or lactating women
* Having given birth in the last year or planning a pregnancy in the next 6 months
* Menopause (as defined by FSH levels ≥30 IU/l)
* Disorders associated with androgen excess and/or menstrual irregularities except PCOS (overt thyroid dysfunction, hyperprolactinemia, adrenal hyperplasia, androgen secreting tumors)
* Malabsorption syndrome
* Intake of medication influencing metabolic or endocrine parameters (insulin sensitizers, oral contraceptives, …), obesity pharmacotherapeutic agents, or calcium supplements in the last 3 months before study entry
* Regular intake of calcium supplements in the last 3 months before study entry
* Lifestyle changes (changes in physical activity) or weight reduction (≥10% of body weight) in the last 3 months before study entry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
fat mass | 12 weeks
  Changes in body fat mass assessed via dual-energy X-ray absorptiometry (DXA) (baseline vs. 12 weeks).

SECONDARY OUTCOMES:
Body weight | 12 weeks
  body weight [kg]
BMI | 12 weeks
  BMI [kg/m²]
waist circumference | 12 weeks
  waist circumference [cm]
hip circumference | 12 weeks
  hip circumference [cm]
Systolic blood pressure | 12 weeks
  systolic blood pressure [mm Hg]
Diastolic blood pressure | 12 weeks
  diastolic blood pressure [mm Hg]
Body composition-lean mass | 12 weeks
  lean mass [kg]
Body composition-total body fat | 12 weeks
  total body fat ([%]
Body composition-gynoid fat mass | 12 weeks
  gynoid fat mass [kg]
Body composition-android fat mass | 12 weeks
  android fat mass [kg]
AUCglucose | 12 weeks
  Metabolic response during an oral glucose tolerance test (oGTT) as defined by AUCglucose
AUCinsulin | 12 weeks
  Metabolic response during an oral glucose tolerance test (oGTT) as defined by AUCinsulin
HOMA-IR | 12 weeks
  Insulin resistance assessed by homeostatic model assessment-insulin resistance (HOMA-IR)
HOMA-beta | 12 weeks
  insulin sensitivity assessed by HOMA-beta
MATSUDA | 12 weeks
  insulin sensitivity assessed by MATSUDA-index
QUICKI | 12 weeks
  insulin sensitivity assessed by Quantitative Insulin-sensitivity Check Index (QUICKI)
Total cholesterol | 12 weeks
  Total cholesterol [mg/dl]
LDL cholesterol | 12 weeks
  LDL cholesterol [mg/dl]
HDL cholesterol | 12 weeks
  HDL cholesterol [mg/dl]
Triglycerides | 12 weeks
  Triglycerides [mg/dl]
HbA1c | 12 weeks
  HbA1c [mmol/mol]
Total testosterone | 12 weeks
  Total testosterone [nmol/l]
Free testosterone | 12 weeks
  Free testosterone [nmol/l]
Free androgen index | 12 weeks
  FAI (Free androgen index)
androstenedione | 12 weeks
  androstenedione [nmol/l]
DHEAS | 12 weeks
  dehydroepiandrosterone sulfate (DHEAS) [µmol/L]
stool microbiome | 12 weeks
  Composition of the stool microbiome Microbiome analysis will be performed through the following steps: patient collection and provision of a stool specimen, DNA isolation from the specimen, PCR reaction to amplify the selected region of the 16S rRNA gene (only present in bacteria), sequencing of the amplicons using next-generation sequencing technology, bioinformatics processing and analysis of the data using suitable software.
Satiety | 12 weeks
  assessed via visual analogue scale [VAS]: "Satiety", minimum score 0, maximum score 10, higher scores mean a worse outcome.
Food craving | 12 weeks
  assessed via visual analogue scale [VAS]: "Food craving", minimum score 0, maximum score 10, higher scores mean a worse outcome.
Quality of life during weight reduction | 12 weeks
  Quality of life assessed via visual analogue scale [VAS]: "How is your quality of life during weight reduction?", minimum score 0, maximum score 10, higher scores mean a better outcome.
Compliance | 12 weeks
  assessed via visual analogue scale [VAS]: "Compliance", minimum score 0, maximum score 10, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Lerchbaum, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Department of Internal Medicine, Division of Endocrinology and Metabolism, Graz, Austria

IPD SHARING:
Plan to Share IPD: No